CLINICAL TRIAL: NCT02455986
Title: A Randomised Controlled Trial of a Pedometer Based Phased Intervention to Encourage Physical Activity in Schools: A Feasibility Study.
Brief Title: The StepSmart Project: A Pedometer Based Phased Intervention to Encourage Physical Activity in Schools
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Responsible Party: Principal Investigator, Dr Mark Tully, Lecturer, Queen's University, Belfast
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: StepSmart
Record Dates: First submitted 2015-05-21; First posted 2015-05-28 (Estimated); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: Physical Activity; Health Behavior; Competitive Behavior; Incentives
MeSH Terms: conditions — Motor Activity; Health Behavior; Competitive Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): The intervention group includes 150 participants aged 12-14 across three schools. Each participant has been given a Fitbit Zip pedometer to wear for a six month period and enrolled on the StepSmart challenge. Participants within the intervention group will take part in two competitions during this period.
  1. School and team based competition. 27/05/15 - 22/06/15 (8 weeks)
  2. Individually focused competition. 22/06/15 - 26/10/15 (18 weeks)
  Prizes of low monetary value will be given to participants based on competition performance
  Interventions: Behavioral: The StepSmart Challenge
- Control (No Intervention): The control group for the study involves approximately 90 participants aged 12 - 14. across two schools. Participants within the control group will complete the same measures as the intervention group including wearing an actigraph GT3X accelerometer for a seven day period and completing all questionnaires at the same time points as the intervention group.

INTERVENTIONS:
Behavioral: The StepSmart Challenge — A six month pedometer based intervention designed to increase Physical Activity in school children
  Arms: Intervention

SUMMARY:
A school based pedometer competition among Year 9 pupils (12 - 14 years old) to promote physical activity (PA).

DETAILED DESCRIPTION:
The intervention is separated into three main phases.

Phase One: A 10-week school competition using pedometers and a range of non-financial incentives e.g. t-shirts, pens, badges etc. (April - June 2015).

Phase Two: End of school competition but participants will still keep the pedometers. We will set them various challenges over the summer to keep active (July - Oct 2015).

Phase Three: Removal of all extrinsically motivation factors. Focus on PA maintenance.

ELIGIBILITY:
Inclusion Criteria

* aged 12-14 years
* enrolled in participating school

Exclusion Criteria

* Unable to give informed consent
* Presence of an underlying medical conditions
* Already enrolled in a physical activity intervention

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 240 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in physical activity as assessed by Actigraph accelerometer | Baseline, 6 months and 1 year
  Actigraph accelerometer counts per minute and minutes of moderate and vigorous physical activity

SECONDARY OUTCOMES:
Change in mental wellbeing measured by the Warwick Edinburgh Mental Well-being Scale | Baseline, 6 months and 1 year
  Warwick Edinburgh Mental Well-being Scale is a validated, self-report instrument assessing mental wellbeing. Possible scores range from range from 14-70, with higher scores indicating higher mental well-being
Change in social support for physical activity measured by the social support for physical activity scale | Baseline, 6 months and 1 year
  Social support for physical activity scale is a validated 5-item scale. Social support is measured as tghe sum of responses to four sub-scales including parental social support (3 items), parental encouragement (2 items), peer support (3 items), and teacher support (3 items). Each question is answered with a 4-point response format ranging from 1 (hardly ever or never) to 4 (every day).
Change in future orientation and impulsivity measured using 8-item time preference scale | Baseline, 6 months and 1 year
  A previously validated 8-item time preference scale is included. Responses are summed to obtain a a future orientation and impulsivity score. High scores reflect future time orientation and greater impulsivity in decision making.

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Tully, PhD, Principal Investigator — Queen's University, Belfast

REFERENCES:
- [Derived] Corepal R, Best P, O'Neill R, Kee F, Badham J, Dunne L, Miller S, Connolly P, Cupples ME, van Sluijs EMF, Tully MA, Hunter RF. A feasibility study of 'The StepSmart Challenge' to promote physical activity in adolescents. Pilot Feasibility Stud. 2019 Nov 17;5:132. doi: 10.1186/s40814-019-0523-5. eCollection 2019. PMID 31832227
- [Derived] Corepal R, Best P, O'Neill R, Tully MA, Edwards M, Jago R, Miller SJ, Kee F, Hunter RF. Exploring the use of a gamified intervention for encouraging physical activity in adolescents: a qualitative longitudinal study in Northern Ireland. BMJ Open. 2018 Apr 20;8(4):e019663. doi: 10.1136/bmjopen-2017-019663. PMID 29678971
- [Derived] Best P, Badham J, Corepal R, O'Neill RF, Tully MA, Kee F, Hunter RF. Network methods to support user involvement in qualitative data analyses: an introduction to Participatory Theme Elicitation. Trials. 2017 Nov 23;18(1):559. doi: 10.1186/s13063-017-2289-5. PMID 29169378